CLINICAL TRIAL: NCT02922088
Title: European (EU) Multi-Center Registry to Assess Outcomes in Patients Undergoing Coronary Artery Bypass Graft (CABG) Surgery: Treatment of Vascular Conduits With DuraGraft®, a Novel Endothelial Damage Inhibitor [VASC]
Brief Title: EU Multicenter Registry to Assess Outcomes in CABG Patients: Treatment of Vascular Conduits With DuraGraft [VASC]
Acronym: VASC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Somahlution LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 005-01
Record Dates: First submitted 2016-09-07; First posted 2016-10-03 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease
Keywords: Vein Graft Failure; Coronary Artery Bypass Graft Surgery; Vascular Grafts; Saphenous Vein Grafts; Vein Graft Disease; Vein Graft Treatment; Vein Graft Handling
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

INTERVENTIONS:
Device: DuraGraft — DuraGraft is a one-time intraoperative vascular graft treatment designed to prevent graft disease and failure and reduce the clinical complications associated with graft failure.

SUMMARY:
The DuraGraft® Registry is a European registry of patients who have undergone CABG and whose vascular grafts have been treated with DuraGraft. All participating sites will be from countries in Europe. The DuraGraft Registry will collect pre-CABG, intraoperative and post-operative data, major post-CABG cardiovascular adverse events, health economic outcomes and patient reported quality of life over a period of 5 years.

DETAILED DESCRIPTION:
Objectives:

(i) To evaluate the Safety and Performance of DuraGraft®

(ii) To characterize the use of DuraGraft and the outcomes of patients whose vascular grafts were treated with DuraGraft in daily clinical routine

(iii) To further characterize the incidence of MACCE outcomes associated with CABG in patients whose vascular grafts were treated with DuraGraft in daily clinical routine

(iv) To compare the use of DuraGraft among hospitals and practices

(v) To obtain patient reported quality of life information

(vi) To obtain important health economics outcomes

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing isolated CABG procedure or CABG plus aortic or mitral valve surgery with at least one saphenous vein or radial artery grafts
* Patient is ≥18 years of age
* Patient (or a legally authorized representative) is willing and able to provide consent
* DuraGraft is being used for the CABG procedure

Exclusion Criteria:

* Participation in a device study or receiving active drug product in an investigational study within one month prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing isolated CABG procedure or CABG plus aortic or mitral valve surgery
Sampling Method: Non-Probability Sample
Enrollment: 2964 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Cardiac Events (MACE) | Annually up to 5 years post-CABG Surgery
  Rate of Major Adverse Cardiac Events: MACE (a composite of Death, Non-Fatal Myocardial Infarction and Repeat Revascularization. The rate of MACE will be compared to historical controls.

SECONDARY OUTCOMES:
Rate of Major Adverse Cardiac and Cerebrovascular Events (MACCE) | Annually up to 5 years post-CABG Surgery
  Rate of Major Adverse Cardiac and Cerebrovascular Events: MACCE (a composite of Death, No-Fatal Myocardial Infarction, Repeat Revascularization and Stroke)
Rate of Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 1 month post-CABG Surgery
  Rate of Major Adverse Cardiac and Cerebrovascular Events: MACCE (a composite of Death, No-Fatal Myocardial Infarction, Repeat Revascularization and Stroke)
Quality of life (EQ-5D-5L) | Annually up to 5 years post-CABG Surgery
  Quality of life will be measured with EQ-5D-5L (Comprised of 5 questions, each with 5 levels that represent 5 health domains (5D): pain, mood, mobility, self-care and daily activities). This overall self-rated health status will be expressed as an index value.
Health Economics Outcomes | Annually up to 5 years post-CABG Surgery
  Health economic outcome measures will include the following:
  * The number (n) of major adverse cardiac and cerebrovascular events (MACCE) will be obtained.
  * The incidence rate (%) of major adverse cardiac and cerebrovascular events (MACCE) will be obtained
  * For death: the mortality rate (%) will be obtained.
  * For non-fatal myocardial infarction, repeat revascularization and stroke: the total number of affected patients (n) will be obtained.
  * For non-fatal myocardial infarction, repeat revascularization and stroke: the total number of the incidence rate (%) will be obtained.
  These outcome measures will be used to obtain the total cost of healthcare resource utilization costs for the treatment of post-operative cardiovascular events.

CONTACTS AND LOCATIONS:
Overall Officials: Maximillian Emmert, MD, Principal Investigator — University Hospital, Zürich
Locations (36):
- Medical University of Vienna, Vienna, Austria
- Germany (15):
  - RWTH Aachen University, Aachen
  - Charité University of Medicine Berlin, Berlin
  - German Heart Center Berlin, Berlin
  - Cologne University Heart Center, Cologne
  - Herzzentrum Dresden, Dresden
  - University Hospital Essen, Essen
  - Goethe University Hospital Frankfurt, Frankfurt
  - University of Giessen, Giessen
  - Georg August University of Gottingen, Göttingen
  - University Medical Center Schleswig-Holstein, Kiel
  - Heart Center Leipzig, Leipzig
  - University of Lubeck, Lübeck
  - University of Marburg, Marburg
  - German Heart Center Munich, München
  - Helios Clinic Wuppertal Heart Center, Wuppertal
- Ireland (2):
  - Cork University Hospital, Cork
  - Galway University Hospitals, Galway
- European Hospital, Roma, Italy
- Spain (11):
  - Complejo Hospitalario Universitario de Badajoz, Badajoz
  - Cruces University Hospital, Barakaldo
  - Hospital Universitario Puerto del Mar, Cadiz
  - Reina Sofia University Hospital, Córdoba
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Gregorio Maran᷉on, Madrid
  - Ruber International Hospital, Madrid
  - Salamanca University Hospital, Salamanca
  - Hospital Universitario De Santiago De Compostela, Santiago de Compostela
  - H.U. Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
- Switzerland (3):
  - Cardiocentro Ticino, Lugano
  - Herzklinik Hirslanden, Zurich
  - University Hospital of Zurich, Zurich
- Medical Park Hospital, Antalya, Turkey (Türkiye)
- United Kingdom (2):
  - Victoria Blackpool Hospital, Blackpool
  - Golden Jubilee National Hospital (Scotland), Clydebank

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data to be determined. A Registry Advisory Committee (RAC) will be formed to provide overall scientific direction for the Registry. A publications sub-committee, composed of a subset of the RAC is planned. This sub-committee will be responsible for overseeing the review and approval of all presentations and all publications related to the DuraGraft Registry.
Time Frame: February 2025
Access Criteria: To be determined

REFERENCES:
- [Background] Kim FY, Marhefka G, Ruggiero NJ, Adams S, Whellan DJ. Saphenous vein graft disease: review of pathophysiology, prevention, and treatment. Cardiol Rev. 2013 Mar-Apr;21(2):101-9. doi: 10.1097/CRD.0b013e3182736190. PMID 22968180
- [Background] Shukla N, Jeremy JY. Pathophysiology of saphenous vein graft failure: a brief overview of interventions. Curr Opin Pharmacol. 2012 Apr;12(2):114-20. doi: 10.1016/j.coph.2012.01.001. Epub 2012 Feb 8. PMID 22321569
- [Background] Thatte HS, Biswas KS, Najjar SF, Birjiniuk V, Crittenden MD, Michel T, Khuri SF. Multi-photon microscopic evaluation of saphenous vein endothelium and its preservation with a new solution, GALA. Ann Thorac Surg. 2003 Apr;75(4):1145-52; discussion 1152. doi: 10.1016/s0003-4975(02)04705-7. PMID 12683553
- [Derived] Sandner S, Misfeld M, Caliskan E, Boning A, Aramendi J, Salzberg SP, Choi YH, Perrault LP, Tekin I, Cuerpo GP, Lopez-Menendez J, Weltert LP, Bohm J, Krane M, Gonzalez-Santos JM, Tellez JC, Holubec T, Ferrari E, Doros G, Vitarello CJ, Emmert MY; Registry Investigators; European DuraGraft Registry investigators'. Clinical outcomes and quality of life after contemporary isolated coronary bypass grafting: a prospective cohort study. Int J Surg. 2023 Apr 1;109(4):707-715. doi: 10.1097/JS9.0000000000000259. PMID 36912566
- [Derived] Caliskan E, Misfeld M, Sandner S, Boning A, Aramendi J, Salzberg SP, Choi YH, Perrault LP, Tekin I, Cuerpo GP, Lopez-Menendez J, Weltert LP, Bohm J, Krane M, Gonzalez-Santos JM, Tellez JC, Holubec T, Ferrari E, Emmert MY; European DuraGraft Registry investigators. Clinical event rate in patients with and without left main disease undergoing isolated coronary artery bypass grafting: results from the European DuraGraft Registry. Eur J Cardiothorac Surg. 2022 Sep 2;62(4):ezac403. doi: 10.1093/ejcts/ezac403. PMID 35929787
- [Derived] Tekin I, Demir M, Ozdem S. Effect of different storage solutions on oxidative stress in human saphenous vein grafts. J Cardiothorac Surg. 2022 Jan 16;17(1):7. doi: 10.1186/s13019-022-01752-7. PMID 35034655
- [Derived] Caliskan E, Sandner S, Misfeld M, Aramendi J, Salzberg SP, Choi YH, Satishchandran V, Iyer G, Perrault LP, Boning A, Emmert MY. A novel endothelial damage inhibitor for the treatment of vascular conduits in coronary artery bypass grafting: protocol and rationale for the European, multicentre, prospective, observational DuraGraft registry. J Cardiothorac Surg. 2019 Oct 15;14(1):174. doi: 10.1186/s13019-019-1010-z. PMID 31615560